CLINICAL TRIAL: NCT00344019
Title: Effects of Single-Dose Atorvastatin on Peri-Procedural Myonecrosis During Percutaneous Coronary Intervention in Patients With Acute Coronary Syndromes - The NO-MI Study
Brief Title: Effects of Atorvastatin on Myonecrosis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2006P000035
Record Dates: First submitted 2006-06-22; First posted 2006-06-26 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Coronary Disease
Keywords: Acute coronary syndrome; Percutaneous coronary intervention; Peri-procedure myocardial infarction
MeSH Terms: conditions — Coronary Disease; Acute Coronary Syndrome | interventions — Atorvastatin; Mass Screening

STUDY DESIGN:
Intervention Model Description: randomized trial of 80 mg atorvastatin vs. placebo pre PCI
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- atorvastatin 80 mg (Active Comparator): 80 mg atorvastatin on average of 2-4 hours pre angio/PCI for ACS
  Interventions: Drug: Atorvastatin 80mg; Other: Screening
- placebo oral tablet (Placebo Comparator): placebo on average of 2-4 hours pre angio/PCI for ACS
  Interventions: Drug: Placebo Oral Tablet; Other: Screening
- Screening (No Intervention): Patients signed consent if willing to participate. Patients will continue onto randomization if appropriate per inc/exc (i.e. stent placement) otherwise screen fail

INTERVENTIONS:
Drug: Placebo Oral Tablet — placebo pre-PCI for ACS
  Arms: placebo oral tablet
Drug: Atorvastatin 80mg — atorvastatin 80 mg pre-angio/PCI
  Other Names: lipitor
  Arms: atorvastatin 80 mg
Other: Screening — Patients signed consent to be screened for eligibility for randomization to placebo vs. study drug (atorvastatin)
  Arms: atorvastatin 80 mg; placebo oral tablet

SUMMARY:
This study is designed as a prospective, randomized, placebo-controlled, double-blind analysis of atorvastatin 80 mg versus placebo administered on average 4 hours prior to percutaneous coronary intervention [PCI] (at least 2 hours) in patients presenting with unstable angina. Only patients with negative cardiac biomarkers, measured on 2 separate occasions a few hours apart will be eligible for inclusion. Furthermore, patients already on high-dose statin therapy; patients taking any statin within 24 hours prior to the PCI; and patients with contraindications to statins will be excluded from the study. The primary endpoint is a quantitative troponin level at 18-24 hours after PCI. At an enrollment of a total of 150 patients (75 per group), the study is powered to detect a 30% difference in troponin level. Secondary endpoints include elevation of creatine kinase (CK) and CK-MB above the upper limit of normal, change in C-reactive protein (CRP) levels from baseline and thrombolysis in myocardial infarction (TIMI) myocardial perfusion grade. All patients will be started on statin therapy the day after the procedure, as deemed appropriate by their treating physicians.

DETAILED DESCRIPTION:
STUDY OBJECTIVES:

1. The primary endpoint of the study is to evaluate the effects of a single high dose of atorvastatin versus placebo on peri-procedural myonecrosis, as measured by troponin T (TnT), during percutaneous coronary intervention (PCI) in patients presenting with acute coronary syndromes (ACS).
2. Secondary endpoints include the measurements of other biomarkers of myocyte injury (CK, CK-MB) and inflammation (CRP).
3. Other secondary endpoints include the relative angiographic efficacy of atorvastatin versus placebo on the post PCI growth of tissue level perfusion circumference and the post PCI growth of tissue level perfusion brightness using digital subtraction angiography.

METHODS:

I. Selection and Number of Patients

The study subjects are to be selected from those patients presenting to the BIDMC for cardiac catheterization. Eligible patients will be identified in the cardiac catheterization holding area prior to their procedure. After obtaining informed consent, patients will be randomized to a single dose of atorvastatin or placebo, which will be administered in the holding area about 4 hours prior to the procedure. There will be a total of 150 subjects enrolled in the study. There are a total of 2500 PCIs performed at the BIDMC per year, a third of which are for ACS. We anticipate that 30-40% of patients with ACS will be eligible for study participation.

II. Informed Consent

Informed consent will be obtained from all individuals prior to enrolment in the study according to local Internal Review Board guidelines.

III. Pretreatment Data Collection

Baseline clinical data will be recorded at enrolment and will include: Subject's age, sex, weight and height, diabetes, hypertension, smoking status, hypercholesterolemia (including cholesterol levels if available), the presence of coronary or peripheral artery disease and prior history of PCI or coronary artery bypass surgery. Further, all current medications will be recorded. A detailed angina history will be collected from the patient and the medical record looking for evidence of unstable angina as defined by Braunwald.

IV. Medications

A. Study Medication

Patients will be randomly assigned to atorvastatin 80 mg po or placebo in a double-blind fashion. The study medication will be administered immediately after informed consent is obtained and the patient is randomized to a treatment group in the cardiac catheterization holding area. Given the typical waiting time between first presentation in the holding area and PCI in a non-emergent case, it is estimated that the study medication will be administered 4 hours prior to the procedure (minimal time of 2 hours). All patients will receive a single dose of study medication prior to the procedure. After the completion of the procedure, all statin therapy will be withheld until the next day. Eligible patients can then receive statin therapy according to the treating physicians' preferences. All potential adverse reactions to the study medication will be recorded.

B. Concomitant Therapy

Aspirin (325 mg/day) will be administered prior to intervention and during follow-up. Clopidogrel (300 mg or 600 mg bolus followed by 75 mg/day) will be administered post-stent deployment. It is expected that the majority of patients will receive a glycoprotein IIb/IIIa inhibitor during the procedure and for 18 hours thereafter.

V. Procedures

A. Laboratory Tests

At baseline, levels of troponin, CK and CK-MB will be obtained at the time of presentation and immediately prior to PCI. Patients with any of these serum markers above the upper limit of normal will be excluded from the study. Post-procedural enzymes will be obtained 6-8 hours after the procedure and the next morning (18-24 hours after the procedure). Patients with elevated enzymes may undergo further sampling to determine the peak enzyme rise. The peak troponin level obtained from any post-procedural blood draw will be used as the primary endpoint. Furthermore, baseline CRP levels will be obtained prior to PCI and on the next day.

B. Digital Subtraction Angiography

To quantitate the kinetics of dye entry into the myocardium, digital subtraction angiography can be used. Digital subtraction angiography will be performed at end diastole by aligning cineframe images before dye filled the myocardium with the frame in which dye first reached its peak brightness. The spine, ribs, diaphragm and the epicardial artery are then subtracted. A representative region of the myocardium is sampled that is free of overlap by epicardial arterial branches to determine the increase in the gray scale brightness of the myocardium. The circumference of the myocardial blush is measured using a handheld planimeter (Fowler, Inc). The frame count ÷ number of frames per second is used to measure the time elapsed during angiography to quantitate the rate of rise in the growth (cm/sec) and brightness (gray/sec) of myocardial blush. Blush will also be assessed visually using the TIMI myocardial perfusion grade.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be aged 18 or over.
* Patients must provide written informed consent.
* Patients are presenting with unstable angina (defined as new onset chest pain, accelerating chest pain, chest pain at rest and ST-segment depression on the electrocardiogram [EKG])
* Patients undergoing successful coronary stent implantation of the (presumed) culprit lesion (defined as < 50% residual stenosis).

Exclusion Criteria:

* Any patient who is unable to give written informed consent.
* Any condition which, in the investigator's opinion, would interfere with optimal participation in the study or produce a significant risk to the patient.
* Patients presenting with an ST-elevation myocardial infarction (MI).
* Patients with elevated troponin, CK, or CK-MB (above the upper limit of normal).
* Patients already on high-dose statin therapy (defined as any statin equivalent to atorvastatin ≥ 40 mg).
* Patients who took any statin agent within 24 hours of presentation to the cardiac catheterization laboratory.
* Patients with active hepatic disease or myositis, in whom statin therapy is contraindicated.
* Patients with hypersensitivity to atorvastatin.
* Patients with procedural complications, including unsuccessful percutaneous transluminal coronary angioplasty (PTCA)/stenting, major side-branch occlusion, flow-limiting dissections at the completion of the procedure, emergent coronary artery bypass surgery, peri-procedural thrombus formation with distal embolization, stent thrombosis within the first 24 hours, repeat emergent PCI within 24 hours, and death within 24 hours.
* Cardiogenic shock.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2006-05 (Actual); Primary Completion 2008-10 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Carrozza, Jr, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
no plans to share data

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients presenting to cath lab for angiogram with unstable angina were approached for participation. If patients agreed to participate, blood was drawn for laboratory evaluation of cardiac enzymes. If enzymes elevated, patient unable to continue participation. Patients proceeded to angiogram as planned. If no PCI performed, patient excluded.
Pre-assignment Details: 97 patients were consented to participate but 74 of them were screen failed afterward due to not meeting angiographic, laboratory or other inclusion criteria. Hence, patients who were screened, but did not complete the study, were not considered enrolled
Groups:
- Screening: Patients that signed consent to participate. Of 97 patients that consented, only 23 completed the study. 74 patients did not continue likely due to no PCI indicated at time of angiogram. Individual subject data no longer available.
Period: Overall Study
Arm/Group | Atorvastatin 80 mg | Placebo Oral Tablet | Screening
Started | 12 | 11 | 74
Completed | 12 | 11 | 0
Not Completed | 0 | 0 | 74
Not completed — did not meet final inclusion criteria | 0 | 0 | 74

BASELINE CHARACTERISTICS:
Population: Study terminated by previous investigator due to slow enrollment. Database no longer available. Data report based on IRB termination report; only gender, race data avail. 97 screened, 23 reported as completed study. Screening data as avail reported herein.
Groups:
- Screening: # patients who signed consent form prior to angiography. 74 did not continue, 23 completed the study. It is believed that most of the 74 did not continue due to the fact that no PCI was indicated at time of angiography
- Total: Total of all reporting groups
Arm/Group | Atorvastatin 80 mg | Placebo Oral Tablet | Screening | Total
Number analyzed (Participants) | 0 | 0 | 97 | 97
Age, Customized [Count of Participants; unit: Participants]
  Age >18 yrs | 0 | 0 | 97 | 97
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  |  | 23 | 23
  Male |  |  | 74 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  |  | 1 | 1
  Not Hispanic or Latino |  |  | 96 | 96
  Unknown or Not Reported |  |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  |  | 0 | 0
  Asian |  |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  |  | 0 | 0
  Black or African American |  |  | 5 | 5
  White |  |  | 85 | 85
  More than one race |  |  | 0 | 0
  Unknown or Not Reported |  |  | 7 | 7
Region of Enrollment [Number; unit: participants]
  United States |  |  | 97 | 97

OUTCOME MEASURES:

1. Primary Outcome: Peri-procedural Myonecrosis
Description: As measured by troponin T (TnT), during percutaneous coronary intervention (PCI). TnT will be measured at 18-24 hours. Assuming a 40% event rate (elevation in TnT), this study powered to predict 30% relative reduction in TnT
Time Frame: 24 hours
Population: Study closed due to slow recruitment and data was not analyzed. Collected data is no longer available as retention period has passed and investigator has left the institution.
Arm/Group | Atorvastatin 80 mg | Placebo Oral Tablet
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Other Biomarkers of Myocyte Injury (CK, CK-MB)
Description: No data was analyzed due to small numbers. Collected data no longer available as retention period has passed
Time Frame: 24 hours
Arm/Group | Atorvastatin 80 mg | Placebo Oral Tablet | Screening
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Inflammatory Markers (CRP)
Description: No data was analyzed due to small numbers. Collected data no longer available as retention period has passed
Time Frame: 24 hours
Arm/Group | Atorvastatin 80 mg | Placebo Oral Tablet | Screening
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Post PCI Growth of Tissue Level Perfusion Circumference and Brightness Using Digital Subtraction Angiography
Description: No data was analyzed due to small numbers. Collected data no longer available as retention period has passed
Time Frame: 24 hours
Arm/Group | Atorvastatin 80 mg | Placebo Oral Tablet | Screening
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Screening: 97 patients screened 23 patients completed study in 1:1 randomization scheme. Randomization assignment not known. Data no longer available. No data analyzed
Arm/Group | Atorvastatin 80 mg | Placebo Oral Tablet | Screening
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 2/97
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 4/97
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin 80 mg (N=0) | Placebo Oral Tablet (N=0) | Screening (N=97)
staged revasculalrization (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — patient readmitted for staged coronary revascularization
increasing shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — patient admitted with increased shortness of breath. ruled out for cardiac cause. pulmonary evaluated. pt discharged home with outpatient follow up scheduled and plans for full pulmonary eval
intracranial hemmorhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — ICH occurred one day post clinically indicated PCI. Patient's family made comfort measures and patient expired
cardiorespiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — patient found pale and non-responsive with HR 40. pt with DNR/DNI status and expired

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No